205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

| | Statistical Arialysis Flatt Fillal |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| <b>Detailed Title:</b> | A phase IV, open-label, single-center study to evaluate |
| | long term immunogenicity up to 15 years after the first |
| | booster immunization with Encepur Adults |
| | (Polygeline-free Tick-borne Encephalitis vaccine for |
| | adults) in adults who received 1 of 3 different primary |
| | vaccination schedules. |
| eTrack study number and | 205847 (TBEV POLYGELINE FREE-025 EXT:021) |
| Abbreviated Title | |
| Scope: | All data pertaining to the above study. |
| <b>Date of Statistical Analysis</b> | Final: 04-Sep-2017 |
| Plan | |
| Co-ordinating author: | PPD |
| Reviewed by: | (Clinical and Epidemiology Project |
| | Lead) |
| | (Clinical Research and Development |
| | Lead) |
| | PPD (Lead statistician) |
| | PPD (Lead statistical analyst) |
| | PPD (Scientific writer) |
| | PPD (Regulatory Affair) |
| | PPD (SERM physician) |
| | (Public disclosure representative) |
| Approved by: | PPD (Clinical and Epidemiology Project |
| | Lead) |
| | PPD (Lead statistician) |
| | PPD (Lead Scientific writer) |
| | (Lead statistical analyst) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 01 April 2017)

# 205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

# **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| LIS | T OF AB | BREVIA | TIONS | | 5 |
| 1. | DOCUN | MENT HI | STORY | | 6 |
| 2. | STUDY | DESIGN | J | | 6 |
| 3. | 3.1. | Primary o | objective | | 8 |
| 4. | 4.1. | Primary I | Endpoints . | ts | 9 |
| 5. | 5.1.<br>5.2. | Definition | n<br>or eliminati | ng data from Analysis Sets | 10 |
| | | 5.2.1.<br>5.2.2. | Elimination 5.2.2.1. 5.2.2.2. 5.2.2.3. | Right censored Data | 11<br>11<br>12 |
| | | | t protocol d | leviation not leading to elimination from per- | |
| 6. | 6.1. | | phy | f demographics/baseline characteristics planned | 12 |
| | | 6.1.2. | in the prot<br>Additional | ocolconsiderations | 12<br>12<br>12 |
| | | 6.2.1.<br>6.2.2.<br>6.2.3.<br>6.2.4.<br>6.2.5. | Additional<br>Efficacy/E<br>Analysis o | f exposure planned in the protocol considerations | 13<br>13 |
| | 6.3. | | genicity<br>Analysis o | f immunogenicity planned in the protocol | 13<br>13 |
| | 6.4. | | of safety<br>Analysis o | f safety planned in the protocol<br>considerations<br>Exclusion of implausible solicited Adverse | 15<br>15<br>16 |
| | | | 6.4.2.2.<br>6.4.2.3.<br>6.4.2.4. | Event | 16<br>16 |
| | | | 6.4.2.5. | Events | |

# 205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

| | Ctatiotical / that y | Jio i iaii i iiiai |
|---|---|---|
| | 6.4.2.6. Concomitant Medication | 17 |
| 7. | ANALYSIS INTERPRETATION | 17 |
| 8. | CONDUCT OF ANALYSES | 18 |
| 9. | CHANGES FROM PLANNED ANALYSES | 18 |
| 10. | LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES | 19 |
| 11. | ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS | 19 |
| | 11.2. Standard data derivation | |

# 205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

# **LIST OF FIGURES**

| | | PAGE |
|---|---|---|
| Figure 1 | Study design of Studies V48P7 | 6 |
| Figure 2 | Study design of study V48P7E1 and TBEV Polygeline-free-023 Ext:021 (V48P7E2) | 7 |
| Figure 3 | Study design of TBEV Polygeline-free-025 Ext:021 | 7 |

# 205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

#### LIST OF ABBREVIATIONS

AE Adverse event

AESI Adverse Events of Special Interest

ANCOVA Analysis of Covariance
ANOVA Analysis of Variance
CI Confidence Interval

eCRF Electronic Case Report Form

CSR Clinical Study Report

CTRS Clinical Trial Registry Summary

EL.U/ml ELISA unit per milliliter

Eli Type Internal GSK database code for type of elimination code

ELISA Enzyme-linked immunosorbent assay

ES Exposed Set

FAS Full Analysis Set

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

GSK GlaxoSmithKline

IU/ml International units per milliliter

LL Lower Limit of the confidence interval

MedDRA Medical Dictionary for Regulatory Activities

N.A. Not ApplicableNT Neutralization testPD Protocol DeviationPPS Per Protocol Set

SAE Serious adverse event SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SUSAR Suspected Unexpected Serious Adverse Reactions

TBE Tick-borne Encephalitis

TBEV Tick-borne Encephalitis virus
TFL Tables Figures and Listings

TOC Table of Content

UL Upper Limit of the confidence interval

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

## 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|---------------------|
| 04-SEP-2017 | Final version | Final – 25-AUG-2017 |

# 2. STUDY DESIGN

The study design of the current study along with the past 2 studies (primary and booster) is presented in the figures below. Figure 1 presents the primary study, Figure 2 presents booster study and Figure 3 presents the current long term follow-up study.

Figure 1 Study design of Studies V48P7



Study V48P7 (205332)

C = Conventional schedule; R = Rapid schedule; AC = Accelerated Conventional schedule; MC = Modified Conventional schedule; Rando = randomisation; LV = Last Visit; V = Visit; D = Day; VAC1, VAC2, VAC3 = vaccination 1, 2 or 3 (indicated in grey);

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

Figure 2 Study design of study V48P7E1 and TBEV Polygeline-free-023 Ext:021 (V48P7E2)



TBE\_R\_B = R-schedule in V48P7 and Booster before enrollment in V48P7E1; TBE\_R = R-schedule in V48P7 and Booster in V48P7E1; TBE\_C = C-schedule in V48P7 and Booster in V48P7E1; TBE\_AC = AC-schedule in V48P7 and Booster in V48P7E1; TBE\_MC = MC-schedule in V48P7 and Booster in V48P7E1; C = Conventional schedule in study V48P7; R = Rapid schedule study V48P7; AC = Accelerated Conventional schedule study V48P7; Enrol = Enrolment; LV = Last Visit; V = Visit; D = Day; Y = Year; BVAC = Booster Vaccination; BS = Blood Sample

Figure 3 Study design of TBEV Polygeline-free-025 Ext:021



TBEV POLYGELINE FREE-025 EXT:021 (205847)

<sup>\*</sup>Booster vaccination 3 years after primary vaccination in V48P7, except TBE R-B (vaccination before enrolment in V48P7E1 and BS only on Day 0)

<sup>\*\*</sup>Study group MC was not followed, it is not a registered schedule; \*\*\*last V48P7E1 visit is screening visit

C = Conventional schedule in study V48P7; R = Rapid schedule study V48P7; AC = Accelerated Conventional schedule study V48P7; Enrol = Enrolment; VAC=Vaccination; LV= Last Visit; V = Visit; D = Day; Y = Year; BS = Blood Sample; SF = safety follow-up

<sup>\*</sup> Approximate number of subjects planned for persistency, number of subjects with a NT titre below 10 during the study cannot be estimated.

<sup>\*\*</sup>Some or all of these visits may not be needed, depending on necessary booster vaccination of subjects.

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

Protocol waivers or exemptions are not allowed unless necessary for the management of immediate safety concerns. Therefore, adherence to the study design requirements, including those specified in the outline of study procedures (Section 5.5 of 205847 "TBEV POLYGELINE FREE-025 EXT:021" protocol Amendment 1 Final: 25 August 2017), are essential and required for study conduct.

- Experimental design: Phase IV, open-label, mono-centric study.
- Duration of the study: For each subject, the study will last less than 5 years.
  - Epoch 001: Persistence evaluation starting at Visit 23 (Year 11) and ending at Visit 27 or Visit 27.2.
- Primary completion Date (PCD): Visit 27.
- End of Study (EoS): Last testing results released of samples collected at Visit 27 or Visit 27 2
- Study groups: Same groups as in study TBEV POLYGELINE FREE (V48)-023EXT:021

## 3. OBJECTIVES

# 3.1. Primary objective

• To evaluate the persistence of antibody response to a booster dose of *Encepur Adults* vaccine starting  $\geq 11$  years after the first booster administration and to continue following subjects up to 15 years after first booster administration.

# 3.2. Secondary objectives

- To evaluate the immune response at 21 days after the second booster dose (boostability) in subjects with an NT titre below 10.
- To evaluate the safety of a second booster dose with regard to SAEs collected after vaccination until study end.

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

## 4. ENDPOINTS

# 4.1. Primary Endpoints

The immunogenicity endpoints will be based on the TBE NT antibody levels in serum at year 11, 12, 13, 14 and 15 as measured by GSK Biologicals' NT.

Measures of immunogenicity are:

- Percentages of subjects with detectable TBE Neutralizing Antibody Titres  $\geq 2$  and  $\geq 10$  as measured by GSK Biologicals' NT.
- Geometric Mean Antibody Titres as measured by GSK Biologicals' NT calculated for each of the different schedule groups.

Endpoints will be summarized according to the immunization schedule received in the V48P7 study and further detailed by the following age subgroups: 25 to 49 years,  $\geq$  50 years and  $\geq$  60 years.

# 4.2. Secondary Endpoints

The immunogenicity endpoints for subjects who received a second booster vaccination will be based on the TBE NT antibody levels in serum at 21 days after the booster vaccination as measured by GSK Biologicals' NT.

Measures of immunogenicity are:

- Percentages of subjects with detectable TBE Neutralizing Antibody Titres ≥ 2 and ≥ 10 as measured by GSK Biologicals' NT, overall and by study group.
- Geometric Mean Antibody Titres and Geometric Mean Ratios (GMRs) blood draw after/before booster as measured by GSK Biologicals' NT, overall and by study group.
- To complement the analysis of persistence, a thorough description of NT waning from year 1 after the first booster dose up to 15 years will be presented for the set of subjects completing the entire 15-year follow-up with no protocol deviations, including those receiving a second booster dose within the previous clinical studies and current study; for those ones, a constant value of NT = 1 from the post booster visit will be used in the analysis. To this end, percentages of subjects with detectable TBE Neutralizing Antibody Titres ≥ 2 and ≥ 10 and GMTs will be presented by study group.

Endpoints will be summarized according to the primary immunization schedule received in the parent study (V48P7).

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

The safety endpoint for subjects who will need a second booster vaccination will be based on SAEs collection after the administration of the booster dose. In vaccinated subjects all SAEs will be collected for 1 month after vaccination. Depending on the timing of the booster dose this will be in the period year 11.5 (Visit 23.1), 12.5 (Visit 24.1), 13.5 (Visit 25.1), or 14.5 (Visit 26.1) or from year 15.5 (Visit 27.1) until 21 days after year 15.5 (Visit 27.2). Post-study SAEs will be collected until study conclusion (Refer Section 8.3.2 of 205847 "TBEV POLYGELINE FREE-025 EXT:021" protocol Amendment 1 Final: 25 August 2017 for details on post-study SAEs)

Measures of safety are:

• Incidence of serious adverse events.

## 5. ANALYSIS SETS

#### 5.1. Definition

Definition of populations:

- a. All Enrolled Population
- all subjects who: have signed an informed consent and have been enrolled
- b. Full Analysis Set-1 (FAS-1)/Modified Intention-to-treat-1 (MITT-1) population, Immunogenicity
- all subjects in the enrolled population who: provide at least one evaluable serum sample
- c. Full Analysis Set-2 (FAS-2)/Modified Intention-to-treat (MITT) population, Immunogenicity
- all subjects in the enrolled population who receive one booster dose during the trial and provide one evaluable serum sample after booster dose
- d. Per Protocol Set/ Per protocol-1 (PP-1) population, Immunogenicity
- all subjects in the FAS-1/MITT-1 Immunogenicity population who: provide evaluable serum samples at the relevant time points and have no major protocol violation as defined in the Statistical Analysis Plan (SAP).
- e. Per Protocol Set/ Per protocol-2 (PP-2) population, Immunogenicity
- all subjects in the FAS-2/MITT-2 Immunogenicity population who: provide evaluable serum samples after booster dose and have no major protocol violation as defined in the Statistical Analysis Plan (SAP).

A major deviation is defined as a protocol deviation that is considered to have a significant impact on the immunogenicity result of the subject.

205847 (TBEV POLYGELINE FREE-025 EXT:021)
Statistical Analysis Plan Final

Examples of major deviations would include:

- confirmed exposure to TBEV (documented diagnosis of TBEV infection) or other Flaviviruses,
- documented TBEV or *Flavivirus* vaccination other than indicated during the course of the study.

The main populations for immunogenicity analyses will be the PPS. FAS will be supplied as sensitivity analyses.

- f. Safety Population
- The safety population will include all subjects who will receive a booster vaccination in this study.

# 5.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each sets.

# 5.2.1. Elimination from Exposed Set (ES)

Not applicable.

# 5.2.2. Elimination from Per-protocol analysis Set (PPS)

## 5.2.2.1. Excluded subjects

A subject will be excluded from the PPS analysis under the following conditions

| Code | Condition under which the code is used |
|---|---|
| 900 | Invalid informed consent or fraud data |
| 150/1040 | Administration of concomitant vaccine(s) forbidden in the protocol |
| 130/1070 | Subjects got vaccinated with the correct vaccine but containing a |
| | lower volume |
| 140/1070 | Vaccination not according to protocol |
| 140/1080 | Vaccine temperature deviation |
| 140/1090 | Expired vaccine administered |
| 200/2010 | Protocol violation (inclusion/exclusion criteria) |
| 230/2040 | Administration of any medication forbidden by the protocol |
| 270/2090 | Subjects did not comply with blood sample schedule |
| 110/2100 | Serological results not available post-vaccination |
| 112/2120 | Obvious incoherence or abnormality or error in data |

Codes referring to vaccination errors or issues are only applicable to those subjects receiving a booster dose at ad-hoc unscheduled visits.

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

## 5.2.2.2. Right censored Data

Not applicable.

## 5.2.2.3. Visit-specific censored Data

Data from visit x will be censored for the PPS analysis under the following conditions.

| Code | Condition under which the code is used |
|---|---|
| 270.x/2090.X | Subjects did not comply with blood sample schedule at visit x |

# 5.3. Important protocol deviation not leading to elimination from per-protocol analysis set

Not applicable.

## 6. STATISTICAL ANALYSES

# 6.1. Demography

# 6.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Descriptive statistics (mean, standard deviation, median, minimum and maximum) for age, height and weight at enrolment will be calculated overall and by vaccine schedule.

Distributions of subjects by sex and ethnic origin will be summarized overall and by vaccine schedule as per parent study assignment.

#### 6.1.2. Additional considerations

In addition to what planned in the protocol, subject distribution by booster visit will be provided per vaccine schedule and overall.

# 6.2. Exposure

Subjects exposed to vaccination will be those who will receive the second booster dose, only if their values go below 10.

## 6.2.1. Analysis of exposure planned in the protocol

Not applicable.

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

#### 6.2.2. Additional considerations

Not applicable.

# 6.2.3. Efficacy/Effectiveness

Not applicable.

## 6.2.4. Analysis of efficacy planned in the protocol

Not applicable.

#### 6.2.5. Additional considerations

Not applicable.

# 6.3. Immunogenicity

# 6.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis population for immunogenicity is the per protocol set and if, in any study group, the percentage of subjects with serological results excluded from the PP set is at least 10%, a second analysis will be performed on the FAS. All analyses entail the calculation of summary statistics by vaccination schedule and age stratification, together with their 95% confidence intervals.

# Long-term immunogenicity (persistence).

- Percentages of subjects with neutralizing antibody titres ≥ 2 and ≥ 10 as measured by NT assay will be tabulated by vaccine schedule (as assigned from the parent study) together with the associated two-sided 95% Clopper-Pearson confidence intervals (CIs). The vaccine schedule difference in the percentage of subjects with neutralizing antibody titres ≥ 2 and ≥ 10 will be calculated using a binomial distribution. The associated confidence interval for these differences will be constructed using the Miettinen-Nurminen method.
- GMTs with the associated 95% CIs will be computed for each vaccine schedule (as assigned from the parent study), by taking the exponential of the corresponding log10-transformed (least squares) means and 95% confidence intervals, from an ANOVA model with group as fixed factor. Vaccine schedule differences along with 95% CIs will also be computed.

SAS code

The SAS statements to calculate the adjusted GMCs will be similar to:

```
PROC glm;
BY vaccinegroup;
CLASS group;
MODEL log_Ab=group;
LSMEANS group / tdiff stderr;
RUN;
```

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

Between-group ratios of GMTs will be calculated by including additional SAS statements within PROC GLM, similar to:

```
ESTIMATE 'Group 1 - Group 2' group 1 -1;
```

Subjects with antibody levels below 10 at a given visit (and that will therefore receive a booster dose) will be kept in the analysis of persistence also for the subsequent years with a value imputed to half of the detection limit, i.e. 1.

Analyses will be conducted on the PPS-1 (and repeated on the FAS-1, if appropriate).

## <u>Immune response to booster dose (boostability):</u>

- Percentages of subjects with neutralizing antibody titres ≥ 2 and ≥ 10 at 21 days after administration of the booster dose, as measured by NT will be tabulated by vaccine schedule (as assigned from the parent study) together with the associated two-sided 95% Clopper-Pearson CIs.
- GMTs with the associated 95% CIs at 21 days after administration of the booster dose, will be computed for each vaccine schedule (as assigned from the parent study), by taking the exponential of the corresponding log10-transformed (least squares) means and 95% confidence intervals, from an ANOVA model with group as fixed factor.

SAS code

The SAS statements to calculate the adjusted GMCs will be similar to:

```
PROC glm;

BY vaccinegroup;

CLASS group;

MODEL log_Ab=group;

LSMEANS group / tdiff stderr;

RUN;
```

Between-group ratios of GMTs will be calculated by including additional SAS statements within PROC GLM, similar to:

```
ESTIMATE 'Group 1 - Group 2' group 1 -1;
```

• GMRs with the associated 95% CIs after/before booster as measured by GSK Biologicals' NT calculated for each of the different schedule groups.

Computationally, the antibody value as recorded prior to the booster visit (i.e. at the previous scheduled clinic visit) will be considered as the denominator for the calculation of the ratio.

Analyses will be conducted on the PPS-2 (and repeated on the FAS-2, if appropriate).

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

#### 6.3.2. Additional considerations

All analyses will be repeated for each age subgroup.

- To complement the analysis of persistence, a thorough description of NT waning from year 1 after the first booster dose up to 15 years will be presented for the set of subjects completing the entire 15-year follow-up with no protocol deviations, including those receiving a second booster dose within the previous clinical studies and current study; for those ones, a constant value of NT = 1 from the post booster visit will be used in the analysis.
- Analysis of boostability will be presented both by time-point (i.e. for each unscheduled visit separately) and aggregated (i.e. all visits considered together).
- Depending on the amount of missing data and as a form of sensitivity analysis, a repeated measure model could be used to evaluate the GMTs persistence.

# 6.4. Analysis of safety

# 6.4.1. Analysis of safety planned in the protocol

In this study, only serious adverse events (SAEs) and pregnancies will be collected.

For vaccinated subjects:

- All pregnancies after vaccination until study end.
- All SAEs will be collected for 1 month after vaccination.
- SAEs leading to study withdrawal

In addition to the above-mentioned reporting requirements and in order to fulfil international reporting obligations, SAEs that are related to study participation (i.e. protocol-mandated procedures, invasive tests, a change from existing therapy) or are related to a concurrent GSK medication/vaccine will be collected and recorded from the time the subject consents to participate in the study until she/he is discharged from the study.

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

An overview of the protocol-required reporting periods for SAEs and pregnancies is given in the table below.

| Event | schedu | led BD | unscheduled V | unscheduled BD | Study |
|---|---|---|---|---|---|
| 0.5 | Visit 23* | Visit 24, 25,<br>26 or 27 | , Visit 23.1, 24.1, 25.<br>or 26.1 | .1 21 days after vaccination<br>visit: Visit 23.2, 24.2, 25.2<br>or 26.2 | conclusion |
| SAEs leading to<br>withdrawal from the<br>study | | | | | |
| SAEs related to | | | | | |
| study participation<br>or concurrent GSK | | | | | |
| medication/vaccine | | | | | |
| SAEs <sup>1</sup> | | | | | |
| Pregnancies <sup>2</sup> | | | | | |

#### 6.4.2. Additional considerations

## 6.4.2.1. Exclusion of implausible solicited Adverse Event

Not applicable.

#### 6.4.2.2. Solicited Adverse Events

Not applicable.

Safety completeness analysis

Not applicable.

## 6.4.2.3. Unsolicited Adverse Events

This analysis applies to all SAEs occurring during the study and related to the study participation or to a concurrent GSK medication/vaccine; additionally, for subjects receiving a booster dose, all SAEs, judged either as probably related, possibly related, or not related to vaccination by the investigator, will be recorded in AE CRF, with a start date on or after the date of booster dose.

<sup>\*</sup>Informed consent obtained before events described below are collected.

V: vaccination; BD: blood draw

<sup>&</sup>lt;sup>1</sup>In vaccinated subjects all SAEs will be collected for 1 month after vaccination.

<sup>&</sup>lt;sup>2</sup> In vaccinated subjects all pregnancies after vaccination until study end

205847 (TBEV POLYGELINE FREE-025 EXT:021)
Statistical Analysis Plan Final

The original verbatim terms used by investigators to identify adverse events in the CRFs will be mapped to preferred terms using the MedDRA dictionary. The serious adverse events will then be grouped by MedDRA preferred terms into frequency tables according to system organ class.

All reported SAEs, as well as SAEs judged by the investigator as at least possibly related to study vaccine, will be summarized according to system organ class and preferred term within system organ class. When an SAE occurs more than once for a subject, the maximal severity and strongest relationship to the vaccine group will be counted.

Separate summaries will be produced for the following categories:

- Serious adverse events.
- Serious adverse events that are possibly or probably related to vaccine.
- Serious Adverse event leading to withdrawal.
- Deaths

Data listings of all serious adverse events and pregnancies will be provided by subject

#### 6.4.2.4. Combined Solicited and Unsolicited Adverse Events

Not applicable.

## 6.4.2.5. Clinical Safety Laboratory Investigations

Not applicable.

#### 6.4.2.6. Concomitant Medication

Medications will be coded using the GSKDRUG dictionary.

The frequencies and percentages of subjects reporting concomitant medications will be tabulated by vaccine schedule and separated for scheduled and unscheduled visit

## 7. ANALYSIS INTERPRETATION

Comparative analyses will be descriptive with the aim to characterise the difference in immunogenicity between groups. No formal statistical comparison will be made.

205847 (TBEV POLYGELINE FREE-025 EXT:021)
Statistical Analysis Plan Final

# 8. CONDUCT OF ANALYSES

# 8.1. Sequence of analyses

Annual listings reporting subjects NT titres will be produced and made available to the investigators. Every year, any subject whose NT titre falls below 10 will be offered a second booster vaccination with *Encepur Adults*.

Final analysis will be conducted after completion of the immunogenicity evaluation at year 15, when the CSR will be produced.

A clinical study report containing all data will be written at study end.

| Description | Analysis<br>ID | Disclosure Purpose (CTRS=public posting, SR=study report, internal) | Dry run<br>review<br>needed<br>(Y/N) | Study Headline Summary (SHS)requiring expedited communication to upper management (Yes/No) | Reference for TFL |
|---|---|---|---|---|---|
| Immunogenicity analysis year 11 | IMM11y | Internal | N | No | 16.2.6.1 |
| Immunogenicity analysis year 12 | IMM12y | Internal | N | No | 16.2.6.1 |
| Immunogenicity analysis year 13 | IMM13y | Internal | N | No | 16.2.6.1 |
| Immunogenicity analysis year 14 | IMM14y | Internal | N | No | 16.2.6.1 |
| Final analysis<br>year 15 | Final | Study report | Y | Yes | All tables and listings in the TOC |

# 8.2. Statistical considerations for interim analysis

The annual evaluations will simply have an informative purpose, evaluating on a yearly basis the subjects who will need a second booster dose. No further statistical considerations need to be applied.

## 9. CHANGES FROM PLANNED ANALYSES

Not applicable.

205847 (TBEV POLYGELINE FREE-025 EXT:021) Statistical Analysis Plan Final

# 10. LIST OF FINAL REPORT TABLES, LISTINGS AND FIGURES

The following group names will be used in the TFLs, to be in line with the T-domains:

| Group order in tables | Group label in tables | Group definition for footnote |
|---|---|---|
| 1 | С | Conventional |
| 2 | R | Rapid |
| 3 | AC | Accelerated Conventional |

The following sub-group names for age class will be used in the TFLs

| Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|
| 1 | 25-49Y | 25-49 years old subjects |
| 2 | >=50Y | >=50 years old subjects |
| 3 | >=60Y | >=60 years old subjects |

# 11. ANNEX 1 STANDARD DATA DERIVATION RULE AND STATISTICAL METHODS

## 11.1. Statistical Method References

The exact two-sided 95% CIs for a proportion within a group will be the Clopper-Pearson exact CI [Clopper CJ, Pearson ES. The use of confidence or fiducial limits illustrated in the case of binomial. *Biometrika*. 1934;26:404-413].

The standardised asymptotic two-sided 95% CI for the group difference in proportions is based on the method described in the following paper:Robert G. Newcombe, interval estimation for the difference between independent proportions: comparison of eleven methods, *Statist Med.* 1998; 17, 873-890]. The standardised asymptotic method used is the method six.

## 11.2. Standard data derivation

#### **NV** legacy

The incomplete date derivations are as follow for an event with start and stop date:

For an incomplete start date, if the day is missing while the month and year are available:

- when the month and year are identical to a complete stop date then the start date is imputed to the stop date.
- when the month and year are not identical to a complete stop date then the start day is imputed to the first day of the month.

205847 (TBEV POLYGELINE FREE-025 EXT:021)
Statistical Analysis Plan Final

For an incomplete start date, if the day and month are missing while the year is available:

- when the year is identical to a complete stop date then the start date is imputed to the stop date.
- when the year is not identical to a complete stop date then the start day/month is imputed to 01Jan.

For an incomplete stop date, if the day is missing while the month and year are available:

- when the month and year are identical to a complete start date then the stop date is imputed to the start date.
- when the month and year are not identical to a complete start date then the stop day is imputed to the first day of the month.

For an incomplete stop date, if the day and month are missing while the year is available:

- when the year is identical to a complete start date then the stop date is imputed to the start date.
- when the year is not identical to a complete start date then the start day/month is imputed to 31dec.